CLINICAL TRIAL: NCT05066321
Title: A Pilot Single Arm Intervention Study of Mindfulness Oriented Recovery Enhancement in Hospitalized People With Opioid Use Disorder
Brief Title: Mindfulness Oriented Recovery Enhancement in Hospitalized People With Opioid Use Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study suspended due to lack of subsequent funding to support the work.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Benjamin Bearnot, M.D., Instructor of Medicine, Department of Medicine, Harvard Medical School; Assistant in Medicine, Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002738
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Opioid-use Disorder
Keywords: Mindfulness; Behavior; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Behavior; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness Oriented Recovery Enhancement (MORE) Arm (Experimental): During hospitalization, participants will receive brief mindfulness training individually in person and complete a series of quantitative baseline questionnaires. Participants will complete 1 MORE session weekly for 8 sessions delivered in small groups of up to 10 people. These sessions will be delivered by a social worker in-person at baseline, and via telehealth after discharge. Follow-up surveys will be conducted at 3-, 6-. 9-, and 12- weeks, and an audio-recorded qualitative exit interview (45-60 minutes) will be completed upon completion of the intervention and the 12-week follow-up survey.
  Interventions: Behavioral: Mindfulness Oriented Recovery Enhancement Sessions

INTERVENTIONS:
Behavioral: Mindfulness Oriented Recovery Enhancement Sessions — The MORE intervention will involve 8 weekly sessions (approximately 1 hour each), during which participants will be taught how to use mindfulness skills to regulate addiction severity, pain, and stress.

SUMMARY:
In this pilot single-armed open-label intervention study of up to 20 individuals with moderate to severe Opioid Use Disorder (OUD)organized into two consecutive groups of up to 10 individuals each, the investigators will measure addiction outcomes and the acceptability and feasibility of adding Mindfulness Oriented Recovery Enhancement (MORE), a promising mind-body therapy to gold standard in-hospital addiction consultation among hospitalized individuals with OUD in advance of a planned two-arm pilot randomized controlled trial.

DETAILED DESCRIPTION:
The investigators will conduct a pilot single-arm intervention study of up to 20 people with moderate to severe OUD. Participants will be enrolled during a hospitalization and receive brief mindfulness training individually in person in the hospital and 8 subsequent sessions of Mindfulness-Oriented Recovery Enhancement (MORE) delivered in small groups of up to 10 people. The intervention will consist of an in-person brief mindfulness training prior to discharge from Massachusetts General Hospital and 8 one-hour group MORE trainings sessions delivered live by a trained addiction social worker over a Zoom telehealth platform.

This study will achieve 2 specific aims. Aim 1 is to quantitatively assess addiction severity, pain, and psychological distress over 12 weeks among people with opioid use disorder receiving manualized Mindfulness-Oriented Recovery Enhancement (MORE) mind-body therapy. Hypothesis 1 is that the receipt of MORE will be associated with decreased addiction severity, pain, and psychological distress among enrolled participants at the end of 12 weeks. Aim 2 is to assess the feasibility and acceptability of conducting a pilot RCT of MORE delivered to people with opioid use disorder and serious bacterial infections. Hypothesis 2 is that more than 50% percent of eligible patients will enroll in the study.

A trained clinical research coordinator (CRC) will attend Addiction Consult Team (ACT) rounds 3 days per week to identify eligible inpatients for this study. Study staff will screen electronic health records (EHR) to confirm eligibility and ask a member of ACT clinical team about the person's suitability to participate given that exclusion criterion may not be known given EHR screening and ACT rounds alone. If the ACT clinician agrees that the participant meets all of the inclusion criteria and none of the exclusion criteria, the ACT clinician will provide the patient with an information sheet about the study. The ACT clinician will then inform the study CRC that the patient has received a brief introduction to the study and is ready to be approached in the hospital using COVID-19 compliant procedures to initiate the consent process.

Prior to receiving the brief mindfulness intervention, enrolled participants will receive and complete a series of quantitative baseline questionnaires (e.g., demographic and substance use history, treatment history) administered by the CRC. These visits will take place in the patient's hospital room (or another private room on the patient's floor in the hospital). At this time, the CRC will also conduct a semi-structured, audio-recorded, qualitative interview with participants. Study outcomes will be assessed in-person at baseline and via mobile phone at 3-, 6-, 9- and 12-week follow-up time points. Upon completion of the intervention and the 12-week follow-up surveys, participants will be asked to complete a 45-60 minute individual exit interview. Informed by an embedded contextual mixed-methods approach, the investigators will also conduct qualitative interviews to better understand why, how, and under what circumstances participants may have achieved reductions in addiction severity in response to MORE.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years old and older
* English-speaking
* Hospitalized at Massachusetts General Hospital, being evaluated by the Addiction Consult Team
* Meet DSM-5 criteria for moderate or severe OUD as documented by Addiction Consult Team

Exclusion Criteria:

* Individuals currently admitted to an Intensive Care Unit
* Individuals who are in legal custody or will not be discharged from a controlled environment during the study period
* Inability to provide informed consent as assessed by the medical team
* Active COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Addiction Severity | 3 months
  The Treatment Effectiveness Assessment, a 4 question validated patient-reported outcome measure, will be used to quantitatively assess recovery from addiction
Enrollment feasibility as measured by the number of individuals who enroll in the study as compared to those who are eligible to enroll | 3 months
  Enrollment percentage as measured by the number of individuals who enroll in the study as compared to those who are eligible to enroll

SECONDARY OUTCOMES:
Distress Tolerance | 3 months
  The Distress Tolerance Scale, a 15 item validated patient-reported outcome measure, will be used to quantitatively assess multiple domains of distress tolerance. The scale ranges from 1 ("strongly agree") to 5 ("strongly disagree"). A higher score indicates a better outcome, with only one item being reverse coded.
Pain Interference | 3 months
  The Patient-Reported Outcome Measurement Information System (PROMIS) Pain Interference scale, a 6 question validated patient-reported outcome measure, will be used to quantitatively assess pain interference. The scale ranges from 1 ("not at all") to 5 ("very much"). A lower score indicates a better outcome.
Pain Severity | 3 months
  The Patient-Reported Outcome Measurement Information System (PROMIS) Pain Severity scale, a 3 question validated patient-reported outcome measure, will be used to quantitatively assess pain severity. The scale ranges from 1 ("had no pain") to 5 ("very severe"). A lower score indicates a better outcome.
Completion of 12-week Follow-up Feasibility | 3 months
  Percentage of those enrolled in the study who complete their 12-week follow-up survey. 100% would be the maximum percentage, and a higher percentage indicates a better outcome.
Completion of at least 4 MORE sessions feasibility | 3 months
  Percentage of those enrolled in the study who complete at least half the MORE sessions

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bearnot, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Division of General Internal Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No